CLINICAL TRIAL: NCT00034515
Title: Ph 1b/2a Study to Assess Levels of INS37217 and Placebo Treatment With Maximum Tolerated Dose Administered by Inhalation Via the Pari LC Star Nebulizer in Adult and Pediatric CF Patients
Brief Title: A Study in Adult and Pediatric Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-102
Record Dates: First submitted 2002-04-29; First posted 2002-04-30 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — denufosol tetrasodium

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Inhalation Solution

SUMMARY:
The purpose of this ascending dose group study is to assess the safety, tolerability, and effects of multiple dose levels of INS37217 and placebo followed by five days twice daily treatment with maximum tolerated dose administered by inhalation via the Pari LC Star nebulizer in adult and pediatric patients with cystic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* FEV1 40-70% (adults)
* FEV1 >/=50% (pediatrics)
* oxygen saturation >90%
* clinically stable
* willing to stay overnight

Exclusion Criteria:

* abnormal renal or liver function
* receiving corticosteroids exceeding 10mg/day or 20 mg every other day
* received intravenous or aerosolized antibiotics 1 week prior to dosing

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2001-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
assess safety and tolerability

SECONDARY OUTCOMES:
assess effects of INS37217 on sputum weight and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director

REFERENCES:
- [Result] Deterding R, Retsch-Bogart G, Milgram L, Gibson R, Daines C, Zeitlin PL, Milla C, Marshall B, Lavange L, Engels J, Mathews D, Gorden J, Schaberg A, Williams J, Ramsey B; Cystic Fibrosis Foundation Therapeutics Development Network. Safety and tolerability of denufosol tetrasodium inhalation solution, a novel P2Y2 receptor agonist: results of a phase 1/phase 2 multicenter study in mild to moderate cystic fibrosis. Pediatr Pulmonol. 2005 Apr;39(4):339-48. doi: 10.1002/ppul.20192. PMID 15704203